CLINICAL TRIAL: NCT00403936
Title: Effects of OA Decompression on Activity of the Autonomic Nervous System
Brief Title: Effects of OA Decompression on the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OAdecompress1
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Muscle Tension
Keywords: osteopathic manipulation; autonomic nervous system

INTERVENTIONS:
Procedure: OA decompression manipulation

SUMMARY:
This study was designed to determine whether a simple manipulative technique of relaxing the tissues of the occipito-atlantal junction in the neck had any effect on the activity of the sympathetic or parasympathetic nervous system. Subjects were dark adapted then measures of pupillary activity, reflecting autonomic nervous system activity were taken before and after treatment. The study hypothesis was that thet treatment technique would have no effect on the pupillary measures, hence indicating no effect on autonomic system activity.

DETAILED DESCRIPTION:
This study was a within subjects/crossover design in which each subject received the treatment and served as his/her own control. 100 subjects were recruited from the student/staff population of the university, were 18 y/o or older with no condition affecting pupillary activity. Pupillary activity was measured with a PLR100 pupillometer and included pupillary diameter, pupillary response latency, maximum constriction velocity and maximum redilation velocity. Subjects were adapted to a dim light environment, measures taken, treatment given at either third or fourth time period and measures retaken. The study was approved by the NSU IRB. Subject numbers were sufficient to have statistical power to find an effect. The study found an effect of treatment on maximum size, showing a decrease with treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o
* Normal accommodation and pupillary response
* Willing to undergo osteopathic manipulation

Exclusion Criteria:

* Active ocular or systemic disease
* Neurologic disease that would alter pupillary response
* Chronic pain syndromes of head or neck
* Pregnant
* Brain injury
* Taking medications that would alter autonomic tone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-04; Study Completion 2005-05

PRIMARY OUTCOMES:
pupillary diameter
pupillary latency
pupillary constriction velocity
pupillary redilation velocity

CONTACTS AND LOCATIONS:
Overall Officials: Chris Piromalli, MSIII, Principal Investigator — College of Osteo Med, Nova Southeastern Univ
Locations (1):
- College of Osteopathic Med, Nova Southeastern Univ, Fort Lauderdale, Florida, United States